CLINICAL TRIAL: NCT06293833
Title: Feasibility Study of Lung Cancer Screening in the Flemish Region, the ZORALCS Study
Brief Title: Implementation of Lung Cancer Screening in the First Line Zone of ZORA (Flanders), Using a Low Dose CT-scan
Acronym: ZORALCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Belgian Cancer Registry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 003315
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer; Smoking Cessation; Lung Cancer, Small Cell
Keywords: Lung Cancer Screening; Lung Cancer; Smoking Cessation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Smoking Cessation; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-risk (ex-) smokers (Experimental): Prevention and early detection of lung cancer are considered the cornerstones to increase the chances of successful treatment and improved outcomes. There is strong scientific evidence that screening for lung cancer through an annual low-dose CT scan (LDCT) in a high-risk population of (ex-)smokers significantly reduces lung cancer mortality and is cost-effective. This implementation study will investigate the participation rate of eligible high risk (ex-)smokers in the First Line Zone (ELZ) South East Region of Antwerp (ZORA) in a LDCT screening program, combined with smoking cessation.
  Interventions: Radiation: Low-dose CT scan; Behavioral: Smoking Cessation

INTERVENTIONS:
Radiation: Low-dose CT scan — Participants get an annual low-dose CT scan in UZA
Behavioral: Smoking Cessation — Smoking cessation campagnes

SUMMARY:
The goal of this clinical trial is to implement lung cancer screening in a targeted high-risk population of heavy (ex-)smokers in Flanders (Belgium). This implementation study will investigate the participation rate of eligible high risk (ex-)smokers in the First Line Zone South East Region of Antwerp (ZORA) in a LDCT screening program, combined with smoking cessation.

DETAILED DESCRIPTION:
A four year prospective non-randomized feasibility implementation study for lung cancer screening in a targeted high-risk population of heavy (ex-)smokers by low-dose CT, combined with a smoking cessation intervention. It will be coordinated by a consortium of researchers from UZA and UAntwerpen.

Lung cancer (LC) remains the leading cause of cancer mortality, worldwide and in Belgium. Prevention and early detection are considered the cornerstones to increase the chances of successful treatment and improved outcomes. There is strong scientific evidence that screening for lung cancer through an annual low-dose CT scan (LDCT) in a high-risk population of (ex-)smokers significantly reduces lung cancer mortality and is cost-effective. This implementation study will investigate the participation rate of eligible high risk (ex-)smokers in the First Line Zone (ELZ) South East Region of Antwerp (ZORA) in a LDCT screening program, combined with smoking cessation. Besides, other indicators of compliance, quality and turn-around-time will be estimated. It will give insights in the feasibility and potential challenges of implementing a LDCT lung cancer screening program in our region. This implementation project is in line with the European Commission Council recommendation of December 2022 to explore the feasibility and effectiveness of LDCT in a high-risk population. Findings from this study will contribute valuable evidence for policymakers and stakeholders. Furthermore, an implementation pilot is a prerequisite for a future high-quality population-based screening program.

ELIGIBILITY:
Inclusion Criteria:

The target population consists of all adult inhabitants from the following municipalities of the ELZ ZORA: Mortsel (2640), Edegem (2650), Boechout (2530), Kontich (2550), Lint (2547), Hove (2540), and having a (TBA) % risk of developing an incidental lung cancer in the following 6 years (calculated a by risk prediction model)

1. Males and females
2. 55 -74 years old
3. Fitness for any kind of curative therapy for lung cancer
4. Absence of prior (lung) cancer in the 5 preceding years (excluding skin basal cell carcinoma and early stage cervical cancer)
5. Having a GP or related trusted health care provider

Exclusion Criteria:

1. participant may not have any symptoms (cough, pain when breathing in...)
2. Body weight >140 kg in view of the maximum charge of the CT-scan table
3. The (rare) hereditary Li-Fraumeni syndrome which gives the carriers an excess risk of X-ray induced oncogenesis

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate of eligible high-risk (ex-)smokers in ELZ-ZORA | 2 years
  Enrollment rate of eligible responders attending at least one LDCT procedure - Measured by descriptive statistics (discrete data)

SECONDARY OUTCOMES:
Responders | 2 years
  Number of candidates responding to the invitation - measured by descriptive statistics (discrete data)
Number of true and false positive nodules | 2 years
  Number of true and false positive nodules detected irequiring further work-up. Measured by descriptive statistics (discrete data)
Impact of smoking cessation intervention | 2 years
  Number of smoking participants having attended a smoking cessation intervention. Measured by descriptive statistics (discrete data)
Success of smoking cessation intervention | 2 years
  Number of smoking participants having quit smoking 1 year after enrollment. Measured by descriptive statistics (discrete data)
Evaluation of shared decision making tool | 2 years
  Evaluation of shared decision making tool by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Snoeckx, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- UZA, Edegem, Antwerp, Belgium